CLINICAL TRIAL: NCT05452980
Title: Sleeve Gastrectomy With Reestablishment of the Acute Angle of His (SG-REACH) in Obese Patients, a Prospective Randomized Controlled Study
Brief Title: Sleeve Gastrectomy With Reestablishment of the Acute Angle of His (SG-REACH) in Obese Patients
Acronym: SG-REACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhen Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG-REACH
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Gastroesophageal Reflux Disease; Excessive Weight Loss; Total Weight Loss; Sleeve Gastrectomy; Angle of His
Keywords: Gastroesophageal Reflux Disease; Sleeve Gastrectomy; Angle of His; Weight Loss
MeSH Terms: conditions — Gastroesophageal Reflux; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleeve gastrectomy (Active Comparator): For standard sleeve gastrectomy (SG), a sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. A security distance of 15 mm lateral to the esophagus is respected to reduce the risk of high leak.
  Interventions: Procedure: sleeve gastrectomy
- SG with reestablishment of the acute angle of His (Experimental): A sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. A security distance of 15 mm lateral to the esophagus is respected to reduce the risk of high leak. Three stitches using nonabsorbable 2-0 Prolone were performed to reestablish the acute angle of His: anterior gastric fundus with esophagus, gastric fundus with left crural diaphragm, posterior gastric fundus with left crural diaphragm.
  Interventions: Procedure: reestablishment of the acute angle of His

INTERVENTIONS:
Procedure: reestablishment of the acute angle of His — A sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. A security distance of 15 mm lateral to the esophagus is respected to reduce the risk of high leak.
  Other Names: sleeve gastrectomy
  Arms: SG with reestablishment of the acute angle of His
Procedure: sleeve gastrectomy — A sleeve was fashioned starting 4 cm proximal to the pylorus using serial applications of an 60 stapler over a 36Fr oro-gastric bougie. A security distance of 15 mm lateral to the esophagus is respected to reduce the risk of high leak.
  Arms: sleeve gastrectomy

SUMMARY:
Gastroesophageal reflux disease (GERD) is one of the most common chronic conditions that can affect one's quality of life. Laparoscopic sleeve gastrectomy (LSG) has become a popular technique and currently is the most frequently practiced surgical operation to treat obesity today. However, the prevalence of GERD following SG can be fairly high. Several studies have noted an incidence between 6% and 47%.

To preserve this natural barrier during SG, a careful dissection at the angle of His must be maintained in order to spare the sling fibers and avoid blunting the angle of His. During creation of the sleeve, the gastric sling fibers are frequently transected near the angle of His, particularly if the transection line is very close to this anatomic landmark. These sling fibers contribute significantly to the function of the LES.

The investigators suggest that after the finishing of SG, the anatomical structure of His horn was destroyed or partly destroyed, and the acute angle of His become obtuse angle. The investigators propose to perform a prospective randomized controlled study to reestablish the acute angle of His in obese patients followig sleeve gastrectomy to prevent GERD.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is one of the most common chronic conditions that can affect one's quality of life. Management of GERD consists primarily in the use of proton pump inhibitors and, in a subset of patients refractory to medical therapy, the use of some form of antireflux surgery. Goals for most antireflux procedures include restoration of a competent lower esophageal sphincter, transhiatal esophageal mobilization to establish 3 cm of intraabdominal esophagus, repair of concomitant hiatus hernia or crura separation, and performance of a partial or total fundoplication. Although the mechanism of action of the surgical fundoplication is multifactorial, one of the most important components is the reestablishment of the acute angle of His through the reconstruction and accentuation of the native musculomucosal, gastroesophageal flap valve.The anatomical mechanisms preventing GERD are the oblique sling fibers of the cardia, the phrenoesophageal ligament, the crura of the diaphragm, and the angle of His. The esophagus normally enters the stomach at an acute angle (the angle of His).

Several factors have been identified including the intrinsic lower oesophageal sphincter (LOS), extrinsic compression of the LOS by the pinchcock action of the crural diaphragm, the length of intra-abdominal oesophagus and the anatomical configuration of the gastric cardia, the angle of His. Emphasis has been placed on either LOS dysfunction, loss of support by the crural diaphragm because of hiatus hernia, or loss of the angle of His. Studies suggested that the angle of His is an important antireflux mechanism. The more acute this angle, the more the gastric fundus will be projected toward the esophagus as gastric distension occurs during a meal. And studies showed that the angle of His plays a role in reflux after distal gastrectomy and that the severity of reflux may be estimated by measuring this angle.

Laparoscopic sleeve gastrectomy (LSG) has become a popular technique and currently is the most frequently practiced surgical operation to treat obesity today. SM-BOSS and SLEEVEPASS studies proved that SG achieve similar weight loss and resolution of obesity-related comorbidities in comparison to those undergoing Roux-en-Y gastric bypass (RYGB). However, the prevalence of GERD following SG can be fairly high. Several studies have noted an incidence between 6% and 47%. This has prompted discussion among the surgical community with regard to the underlying pathomechanisms of GERD after SG and the postoperative management of reflux disease. So far, a number of new techniques have been reported to yield more encouraging results with regard to reflux symptoms after SG, but most evidence originates from retrospective studies with a small number of cases or is based on experts' opinions. The available data are limited, and very heterogeneous.

To preserve this natural barrier during SG, a careful dissection at the angle of His must be maintained in order to spare the sling fibers and avoid blunting the angle of His. During creation of the sleeve, the gastric sling fibers are frequently transected near the angle of His, particularly if the transection line is very close to this anatomic landmark. These sling fibers contribute significantly to the function of the LES.

The investigators suggest that after the finishing of SG, the anatomical structure of His horn was destroyed or partly destroyed, and the acute angle of His become obtuse angle. The investigators propose to perform a prospective randomized controlled study to reestablish the acute angle of His in obese patients followig sleeve gastrectomy to prevent GERD.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 32.5 kg/m2 with or without T2DM;
* 27.5 kg/ m2 < BMI < 32.5 kg/m2 with T2DM but failed conservative treatment and combined with at least two metabolic diseases or comorbidities;
* Duration of T2DM ≤15 years with fasting Cpeptide ≥ 50% of normal lower limit
* Waist circumference: male ≥ 90 cm, female ≥ 85 cm
* Age within 16~65 years old

Exclusion Criteria:

* GERD preoperatively
* Hiatus hernia approved by gastroscopy preoperatively
* Pregnancy;
* A history of mental illness and neurological disease;
* The patient refuses surgery;
* Combined with pituitary tumor;
* Long-term use of antidepressant drugs;
* Long-term use of immunosuppressants;
* Situations in which the investigator or other examiner considers from the enrolled study that there are good reasons for nonconformity: if there are potential inconsistencies with the clinical protocol

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of gastroesophageal reflux disease | 1 year
  The rate of gastroesophageal reflux disease following sleeve gastrectomy at 1 year

SECONDARY OUTCOMES:
Complications | 30 days postoperatively]
  Complications within 30 days postoperatively
Operating time | During the operation
  Time from opeing of the operation to the end of the operation
excessive weight loss | 3 months, 6 months, 1 year, 3 years and 5 years postoperatively
  Percentage of excess weight loss (EWL) at any time postoperative was calculated as the amount of weight loss divided by the amount of excess weight times 100%.
total weight loss | 3 months, 6 months, 1 year, 3 years and 5 years postoperatively
  total weight loss compared with preoperative weight

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jun Wang, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No